CLINICAL TRIAL: NCT01889602
Title: Characterizing and Predicting Drug Effects on Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CPDEC
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Cognitive Deficits
Keywords: Healthy volunteers; Topiramate; Neurocognition; Drug-induced cognitive deficits
MeSH Terms: conditions — Cognition Disorders | interventions — Lorazepam; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Topiramate 100mg (Experimental): Participant will receive 3 single-dose treatments with 2-week washout between each treatment. At each of 3 treatments, participants will receive 100mg torpiramate, 2mg lorazepam, or placebo. Treatment order is randomized. All participants in this arm will receive all 3 treatments.
  Interventions: Drug: Lorazepam; Other: Placebo; Drug: Topiramate 100mg
- Topiramate 150mg (Experimental): Participant will receive 3 single-dose treatments with 2-week washout between each treatment. At each of 3 treatments, participants will receive 150mg torpiramate, 2mg lorazepam, or placebo. Treatment order is randomized. All participants in this arm will receive all 3 treatments.
  Interventions: Drug: Lorazepam; Other: Placebo; Drug: Topiramate 150mg
- Topiramate 200mg (Experimental): Participant will receive 3 single-dose treatments with 2-week washout between each treatment. At each of 3 treatments, participants will receive 200mg torpiramate, 2mg lorazepam, or placebo. Treatment order is randomized. All participants in this arm will receive all 3 treatments.
  Interventions: Drug: Lorazepam; Other: Placebo; Drug: Topiramate 200mg

INTERVENTIONS:
Drug: Lorazepam — Lorazepam: 2mg, po, 1x
  Other Names: Ativan
Other: Placebo — Non-active placebo, po, 1x
Drug: Topiramate 100mg — Topiramate: 100 mg, po, 1x
  Other Names: Topamax
  Arms: Topiramate 100mg
Drug: Topiramate 150mg — Topiramate: 150 mg, po, 1x
  Other Names: Topamax
  Arms: Topiramate 150mg
Drug: Topiramate 200mg — Topiramate: 200 mg, po, 1x
  Other Names: Topamax
  Arms: Topiramate 200mg

SUMMARY:
Cognitive impairment is a widely reported side effect of many commonly used drugs. Even a mild, untoward effect on an essential function such a linguistic behavior, a directly observable product of complex cognitive processes, is disruptive to daily life. Nevertheless, the mechanisms underlying a drug's impact on cognition are poorly understood. This lack of understanding impedes the ability to predict both the effects of drugs in development and the degree to which an individual is vulnerable to the cognitive impact of a particular agent. Topiramate (TPM, an antiepileptic drug) is, with increasing frequency, being prescribed for a range of conditions including migraine prophylaxis, obesity and pain. It is a prime example of a drug that causes speech and language problems severe enough in some patients to result in discontinuation of therapy. For reasons not well understood, TPM has a poorer cognitive profile than many of the older antiepileptic drugs. The investigators' rational for this study is that it will offer insight into the mechanisms underlying drug-induced cognitive deficits.

DETAILED DESCRIPTION:
The investigators' long-term goal is to enhance clinical strategies and inform drug development in order to maximize the benefits of individual drug therapy while minimizing adverse cognitive/language-related side effects. The investigators' objective in this application is to elucidate the relationship among drug exposure as measured by plasma drug levels, its neurophysiological effects, and consequent effects on the cognitive processes observable in everyday language use. Using topiramate (TPM) as a prototype, the investigators will apply the tools of clinical pharmacology, computational linguistics, neuroscience, and engineering to the design and execution of randomized, double blind, crossover studies using three (3) doses of TPM, one (1) dose of a comparator drug (lorazepam-LZP) and a placebo. In order to isolate the cognitive effects of TPM from those possibly arising from an underlying medical condition, subjects will be healthy adults. The investigators will capitalize on an innovative system for automated language and speech analysis (SALSA) developed in our laboratory, to quantify the effects of TPM administration on effective language use, a crucial component of normal day-to-day functioning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Ages 18-50
* Women are post-menopausal or using approved birth control methods
* To control for brain lateralization of language functions, subjects need to have a dominant right hand.

Exclusion Criteria:

* Presence of clinically significant cardiovascular, endocrine, hematopoietic, hepatic, renal, neurologic, and/or psychiatric disease including suicidality
* Vision or hearing impairments
* Current or a history of drug or alcohol abuse
* living outside of the Twin Cities Metropolitan area.
* The use of concomitant medications known to affect Topiramate (TPM), Lorazepam (LZP), or the use of any concomitant medications that may alter cognitive function
* Prior adverse reaction or prior hypersensitivity to TPM, LZP or related compounds
* A positive pregnancy test (administered to all women before enrollment, and prior to each study session).
* Subjects who have received any investigational drug within the previous 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Marino, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Callisto SP, Illamola SM, Birnbaum AK, Barkley CM, Bathena SPR, Leppik IE, Marino SE. Severity of Topiramate-Related Working Memory Impairment Is Modulated by Plasma Concentration and Working Memory Capacity. J Clin Pharmacol. 2020 Sep;60(9):1166-1176. doi: 10.1002/jcph.1611. Epub 2020 Apr 16. PMID 32297992

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate 100mg: Randomized to Topiramate; 100mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
  Topiramate: Topiramate: 100 mg, 150 mg or 200 mg, po, 1x
- Topiramate 150mg: Randomized to Topiramate; 150mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
  Lorazepam: Lorazepam: 2mg, po, 1x
- Topiramate 200mg: Randomized to Topiramate; 200 mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
  Placebo
Period: First Intervention
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 20 | 20 | 20
Completed | 19 | 17 | 18
Not Completed | 1 | 3 | 2
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Study ending | 0 | 1 | 0
Period: First Washout Period of at Least 2 Weeks
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 19 | 17 | 18
Completed | 19 | 17 | 18
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 19 | 17 | 18
Completed | 18 | 17 | 16
Not Completed | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Study ending | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Second Washout Period of at Least 2 Week
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 18 | 17 | 16
Completed | 18 | 17 | 16
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 18 | 17 | 16
Completed | 15 | 15 | 16
Not Completed | 3 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Period: Third Washout Period of at Least 2 Weeks
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg
Started | 15 | 15 | 16
Completed | 15 | 15 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: To address reviewer comments about inconsistencies between participate flow and baseline population: Baseline analysis population is only subjects who completed the trial. The participant flow section is divided into time periods. The baseline characteristics are divided by intervention. The two sections will not correspond.
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg | Total
Number analyzed (Participants) | 14 | 15 | 17 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 17 | 46
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Years] | 31.9 (11.48) | 38.54 (10.21) | 26.41 (8.42) | 28.52 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 6 | 7 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 3 | 12
  White | 8 | 8 | 9 | 25
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 17 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in COWA Unique Word Count
Description: Study has 3 arms (100mg, 150mg, or 200mg topiramate) and 3 periods per arm (topiramate, 2mg lorazepam, or placebo). Topiramate (TPM), Lorazepam (LZP), or Placebo (PLA) was given to the participant at the beginning of Sessions 2, 3, and 4 (crossover design). No drug was given at Sessions 1 and 5. The baseline value was defined as the average of the values at Session 1 and Session 5. The change from baseline for Topiramate is the value at 2.5 hours post-dose at the Topiramate visit minus the value at baseline, divided by the value at baseline; similarly for Lorazepam and Placebo.
Time Frame: Session 1 to Session 5
Measure: Mean (Standard Deviation); unit: Word Count
Groups:
- Arm: Topiramate 100mg, Period: Topiramate: Randomized to Topiramate; 100mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the topiramate period.
  Topiramate: 100 mg po, 1x
- Arm:Topiramate 150mg, Period: Topiramate: Randomized to Topiramate; 150mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the topiramate period.
  Topiramate: 150 mg po, 1x
- Arm: Topiramate 200mg, Period: Topiramate: Randomized to Topiramate; 200mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the topiramate period.
  Topiramate: 200 mg po, 1x
- Arm: Topiramate 100mg, Period: Lorazepam: Randomized to Topiramate; 100mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the lorazepam period.
  Lorazepam: 2 mg po, 1x
- Arm: Topiramate 150mg, Period: Lorazepam: Randomized to Topiramate; 150mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the lorazepam period.
  Lorazepam: 2 mg po, 1x
- Arm: Topiramate 200mg, Period: Lorazepam: Randomized to Topiramate; 200mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the lorazepam period.
  Lorazepam: 2 mg po, 1x
- Arm: Topiramate 100mg, Period: Placebo: Randomized to Topiramate; 100mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the placebo period.
  Placebo: po, 1x
- Arm: Topiramate 150mg, Period: Placebo: Randomized to Topiramate; 150mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the placebo period.
  Placebo: po, 1x
- Arm: Topiramate 200mg, Period: Placebo: Randomized to Topiramate; 200mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments. This is the placebo period.
  Placebo: po, 1x
Arm/Group | Arm: Topiramate 100mg, Period: Topiramate | Arm:Topiramate 150mg, Period: Topiramate | Arm: Topiramate 200mg, Period: Topiramate | Arm: Topiramate 100mg, Period: Lorazepam | Arm: Topiramate 150mg, Period: Lorazepam | Arm: Topiramate 200mg, Period: Lorazepam | Arm: Topiramate 100mg, Period: Placebo | Arm: Topiramate 150mg, Period: Placebo | Arm: Topiramate 200mg, Period: Placebo
Number analyzed (Participants) | 14 | 15 | 17 | 14 | 15 | 17 | 14 | 15 | 17
Word Count | -0.407725385 (0.110593408) | -0.425898667 (0.186240451) | -0.412534118 (0.154640084) | -0.108298333 (0.240452491) | 0.131452143 (0.263967943) | -0.095221176 (0.228163172) | -0.011651538 (0.152526619) | 0.077431333 (0.176020802) | 0.047164706 (0.166162762)

2. Primary Outcome: Change From Baseline in Spontaneous Narrative Raw Word Count
Description: as for outcome 1
Time Frame: Session 1 to Session 5
Measure: Mean (Standard Deviation); unit: Word Count
Arm/Group | Arm: Topiramate 100mg, Period: Topiramate | Arm:Topiramate 150mg, Period: Topiramate | Arm: Topiramate 200mg, Period: Topiramate | Arm: Topiramate 100mg, Period: Lorazepam | Arm: Topiramate 150mg, Period: Lorazepam | Arm: Topiramate 200mg, Period: Lorazepam | Arm: Topiramate 100mg, Period: Placebo | Arm: Topiramate 150mg, Period: Placebo | Arm: Topiramate 200mg, Period: Placebo
Number analyzed (Participants) | 14 | 15 | 17 | 14 | 15 | 17 | 14 | 15 | 17
Word Count | -0.01596 (0.360237984) | -0.131732 (0.192165204) | -0.323135625 (0.297067179) | 0.109636 (0.236323153) | 0.016635385 (0.283748379) | -0.128177333 (0.281246222) | 0.117455385 (0.360519103) | -0.01098 (0.272331286) | 0.011456471 (0.225720885)

ADVERSE EVENTS:
Time Frame: 30 days following the last administration of study drug.
Description: Study is a 3x3 latin square design with 3 arms (100mg, 150mg, or 200mg topiramate) and 3 periods per arm (topiramate, 2mg lorazepam, or placebo). Topiramate (TPM), Lorazepam (LZP), or Placebo (PLA) was given to the participant at the beginning of Sessions 2, 3, and 4 (crossover design). Sessions 1 and 5 are washouts.
Groups:
- Topiramate 100mg: Randomized to Topiramate; 100mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
- Topiramate 150mg: Randomized to Topiramate; 150mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
- Topiramate 200mg: Randomized to Topiramate; 200 mg; lorazepam 2mg or placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
- Lorazepam 2mg: Randomized to Topiramate; 100, 150, or 200 mg; lorazepam 2mg; Each subject in this arm received each treatment in random order with a two-week washout between treatments
- Placebo: Randomized to Topiramate; 100, 150, or 200 mg; placebo; Each subject in this arm received each treatment in random order with a two-week washout between treatments
Arm/Group | Topiramate 100mg | Topiramate 150mg | Topiramate 200mg | Lorazepam 2mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/17 | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/17 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 1/17 | 0/46 | 0/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate 100mg (N=14) | Topiramate 150mg (N=15) | Topiramate 200mg (N=17) | Lorazepam 2mg (N=46) | Placebo (N=46)
Eye Twitching (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT01889602/Prot_SAP_000.pdf